CLINICAL TRIAL: NCT03560440
Title: Evaluation of the Dosing Regimen of Vancomycin in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Isabelle Spriet, PharmD PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56779
Record Dates: First submitted 2016-11-29; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: Vancomycin; Pharmacokinetics; Trough level; Pediatric
MeSH Terms: conditions — Gram-Positive Bacterial Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Plasma exposure vancomycin: Pediatric patients treated with vancomycin
  Interventions: Other: Plasma exposure vancomycin

INTERVENTIONS:
Other: Plasma exposure vancomycin — Investigation of plasma exposure of vancomycin.

SUMMARY:
In this retrospective registry the investigators wish to verify whether the current dosing regime of vancomycin is leading to the appropriate pharmacokinetic targets in pediatric patients. Therefore data will be collected from all pediatric patients hospitalized in University Hospitals Leuven between January 2012 and April 2014 who were treated with vancomycine.

DETAILED DESCRIPTION:
In this retrospective registry the investigators wish to verify whether the current dosing regime of vancomycin is leading to the appropriate pharmacokinetic targets in pediatric patients. Therefore data will be collected from all pediatric patients hospitalized in University Hospitals Leuven between January 2012 and April 2014 who were treated with vancomycine. Patient files will be screened for relevant information. Individual patients can be included multiple times if vancomycin has been administered more than once.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients hospitalized in the University Hospitals Leuven between January 2012 and April 2014, treated with vancomycin

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients treated with vancomycin and hospitalized in UZ Leuven between January 2012 and April 2014
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Loading dose related plasma exposure vancomycin | 24 hours after loading dose
  Plasma exposure to vancomycin in relation to administered dose

OTHER OUTCOMES:
Loading dose related plasma exposure vancomycin | 24 hours after dosage adjustment
  Plasma exposure to vancomycin in relation to administered dose

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rybak MJ, Lomaestro BM, Rotschafer JC, Moellering RC, Craig WA, Billeter M, Dalovisio JR, Levine DP. Vancomycin therapeutic guidelines: a summary of consensus recommendations from the infectious diseases Society of America, the American Society of Health-System Pharmacists, and the Society of Infectious Diseases Pharmacists. Clin Infect Dis. 2009 Aug 1;49(3):325-7. doi: 10.1086/600877. PMID 19569969
- [Background] Piro CC, Crossno CL, Collier A, Ho R, Koyama T, Frangoul H. Initial vancomycin dosing in pediatric oncology and stem cell transplant patients. J Pediatr Hematol Oncol. 2009 Jan;31(1):3-7. doi: 10.1097/MPH.0b013e31818b3520. PMID 19125078
- [Background] Glover ML, Cole E, Wolfsdorf J. Vancomycin dosage requirements among pediatric intensive care unit patients with normal renal function. J Crit Care. 2000 Mar;15(1):1-4. doi: 10.1053/jcrc.2000.0150001. PMID 10757191
- [Background] Kim DI, Im MS, Choi JH, Lee J, Choi EH, Lee HJ. Therapeutic monitoring of vancomycin according to initial dosing regimen in pediatric patients. Korean J Pediatr. 2010 Dec;53(12):1000-5. doi: 10.3345/kjp.2010.53.12.1000. Epub 2010 Dec 31. PMID 21253314
- [Background] Ito H, Shime N, Kosaka T. Pharmacokinetics of glycopeptide antibiotics in children. J Infect Chemother. 2013 Apr;19(2):352-5. doi: 10.1007/s10156-012-0458-8. Epub 2012 Aug 8. PMID 22872188